CLINICAL TRIAL: NCT01095510
Title: Open-Label, Single-Dose Study to Evaluate the Response and Pharmacokinetics/Pharmacodynamics of Different Doses of CINRYZE® [C1 Inhibitor (Human)] For Treatment of Acute Angioedema Attacks in Children Less Than 12 Years of Age With Hereditary Angioedema
Brief Title: CINRYZE for the Treatment of Hereditary Angioedema Attacks in Children Under the Age of 12
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0624-203; 2011-000369-11 (EudraCT Number)
Record Dates: First submitted 2010-03-24; First posted 2010-03-30 (Estimated); Results first posted 2014-07-25 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: CINRYZE; C1 INH; HAE; C1 inhibitor; Pediatric; PK/PD
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — SERPING1 protein, human; Complement C1 Inhibitor Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 500 U CINRYZE (10-25 kg body weight) (Experimental): Single IV dose of 500 U CINRYZE
  Interventions: Biological: CINRYZE
- 1000 U CINRYZE (10-25 kg body weight) (Experimental): Single IV dose of 1000 U CINRYZE
  Interventions: Biological: CINRYZE
- 1000 U CINRYZE (>25 kg body weight) (Experimental): Single IV dose of 1000 U CINRYZE
  Interventions: Biological: CINRYZE
- 1500 U CINRYZE (>25 kg body weight) (Experimental): Single IV dose of 1500 U CINRYZE
  Interventions: Biological: CINRYZE

INTERVENTIONS:
Biological: CINRYZE
  Other Names: C1 inhibitor [human]

SUMMARY:
The objectives of this study were to evaluate: (1) the dose response and (2) the pharmacokinetics (PK) and pharmacodynamics (PD) of intravenous (IV) administration of CINRYZE for the treatment of acute angioedema attacks in children above and below 25 kg and less than 12 years of age with hereditary angioedema (HAE); and (3) to determine the safety and tolerability following IV administration of CINRYZE in this study population.

DETAILED DESCRIPTION:
Each subject received CINRYZE for treatment of a single acute angioedema attack.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this protocol, subjects must:

1. Be at least 10 kg of body weight.
2. Have a confirmed diagnosis of HAE.
3. Have an acute HAE attack and be able to initiate treatment within 8 hours after onset of symptoms.

Exclusion Criteria:

To be eligible for this protocol, subjects must not:

1. Have any active infectious illness.
2. Have had a prior HAE attack and/or received any C1 INH product within 7 days prior to dosing with study drug.
3. Have received therapy with antifibrinolytics (e.g., tranexamic acid), androgens (e.g., danazol, oxandrolone, stanozolol, or testosterone), ecallantide (Kalbitor®), or icatibant (Firazyr®) within 7 days prior to dosing with study drug.
4. Have a history of allergic reaction to C1 INH products, including CINRYZE (or any of the components of CINRYZE), or other blood products.
5. Have participated in any other investigational drug evaluation within 30 days prior to dosing with study drug, or have previously received treatment with CINRYZE in this study at any time.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2010-06-02 (Actual); Primary Completion 2012-04-17 (Actual); Study Completion 2012-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- United States (8):
  - Asthma & Allergy Associates, P.C., Colorado Springs, Colorado
  - University of South Florida Asthma, Allergy and Immunology Clinical Research Unit, Tampa, Florida
  - Institute for Asthma and Allergy, PC, Chevy Chase, Maryland
  - Allergy & Asthma Research Group, Eugene, Oregon
  - Baker Allergy, Asthma and Dermatology Research Center, LLC, Lake Oswego, Oregon
  - AARA Research Center, Dallas, Texas
  - Allergy and Asthma Research Center, P.A., San Antonio, Texas
  - Marycliff Allergy Specialists, Spokane, Washington
- Germany (2):
  - Charité Universitätsmedizin Berlin, Dept. of Dermatology and Allergy, Berlin
  - Klinikum rechts der Isar, Technical University Munich, ENT Clinic, Munich
- Semmelweis University, Allergy and Angioedema Outpatients Clinic, Kútvölgyi Clinical Center, Budapest, Hungary

REFERENCES:
- [Result] Lumry W, Soteres D, Gower R, Jacobson KW, Li HH, Chen H, Schranz J. Safety and efficacy of C1 esterase inhibitor for acute attacks in children with hereditary angioedema. Pediatr Allergy Immunol. 2015 Nov;26(7):674-80. doi: 10.1111/pai.12444. Epub 2015 Aug 11. PMID 26171584

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were not enrolled in the lower body weight category (10-25 kilograms [kg]) 1000 Units (U) dose group despite substantial recruitment efforts.
Pre-assignment Details: Of 12 participants screened, 9 participants were enrolled and treated. The reason for 3 participants were screen failures as they did not meet the inclusion criteria.
Groups:
- 500 U CINRYZE (10-25 kg Body Weight): Single intravenous (IV) dose of 500 U CINRYZE
Period: Overall Study
Arm/Group | 500 U CINRYZE (10-25 kg Body Weight) | 1000 U CINRYZE (10-25 kg Body Weight) | 1000 U CINRYZE (>25 kg Body Weight) | 1500 U CINRYZE (>25 kg Body Weight)
Started | 3 | 0 | 3 | 3
Completed | 3 | 0 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 500 U CINRYZE (10-25 kg Body Weight) | 1000 U CINRYZE (>25 kg Body Weight) | 1500 U CINRYZE (>25 kg Body Weight) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Continuous [Median (Full Range); unit: years] | 7 [6 to 9] | 9 [7 to 9] | 10 [8 to 11] | 9 [6 to 11]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 8
  Male | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Presence of Unequivocal Beginning of Relief of the Defining Attack Symptom
Time Frame: Within 4 hours following treatment
Population: Intent-to-treat efficacy (ITT-E) population included all participants with baseline and at least one post-infusion investigator assessment of the hereditary angioedema (HAE) attack.
Measure: Number; unit: participants
Arm/Group | 500 U CINRYZE (10-25 kg Body Weight) | 1000 U CINRYZE (>25 kg Body Weight) | 1500 U CINRYZE (>25 kg Body Weight)
Number analyzed (Participants) | 3 | 3 | 3
participants
  Yes | 3 | 3 | 3
  No | 0 | 0 | 0

2. Secondary Outcome: Time to Unequivocal Beginning of Relief of the Defining Attack Symptom
Time Frame: Within 4 hours following treatment
Population: ITT-E population
Measure: Median (Full Range); unit: hours
Arm/Group | 500 U CINRYZE (10-25 kg Body Weight) | 1000 U CINRYZE (>25 kg Body Weight) | 1500 U CINRYZE (>25 kg Body Weight)
Number analyzed (Participants) | 3 | 3 | 3
hours | 1.25 [0.25 to 1.75] | 0.25 [0.25 to 0.50] | 0.50 [0.25 to 2.50]

3. Secondary Outcome: Time to Complete Resolution of the Attack
Time Frame: Within 1 week following treatment
Population: ITT-E population.
Measure: Median (Full Range); unit: hours
Arm/Group | 500 U CINRYZE (10-25 kg Body Weight) | 1000 U CINRYZE (>25 kg Body Weight) | 1500 U CINRYZE (>25 kg Body Weight)
Number analyzed (Participants) | 3 | 3 | 3
hours | 13.58 [11.48 to 37.35] | 10.00 [1.57 to 22.33] | 29.07 [1.58 to 102.33]

4. Secondary Outcome: Change in C1 Inhibitor (C1 INH) Antigen and Functional C1 INH Concentrations
Description: Data was not reported due to change in planned analysis.
Time Frame: Pre-dose, 2, 4, 8 hours post dose on Day 1; Day 2, 3, 5, 8
Population: No participant agreed to obtain pharmacokinetic (PK) blood sampling for antigenic and functional C1 INH levels. Hence, it was planned not to be analyzed.
Arm/Group | 500 U CINRYZE (10-25 kg Body Weight) | 1000 U CINRYZE (>25 kg Body Weight) | 1500 U CINRYZE (>25 kg Body Weight)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected through 1 week following the dose of study drug.
Arm/Group | 500 U CINRYZE (10-25 kg Body Weight) | 1000 U CINRYZE (>25 kg Body Weight) | 1500 U CINRYZE (>25 kg Body Weight)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 500 U CINRYZE (10-25 kg Body Weight) (N=3) | 1000 U CINRYZE (>25 kg Body Weight) (N=3) | 1500 U CINRYZE (>25 kg Body Weight) (N=3)
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Change in C1 INH antigen and functional C1 INH concentrations endpoint was not analyzed as no participants agreed to additional and optional blood sampling. As a result, no PK parameters were calculated for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Trial Agreement. Most restrictive provision - PI will not publish results until after first of: multicenter publication is published or 24 months from study end. Thereafter, PI may publish his results. PI must provide copy of proposed publication to Sponsor for pre-review. If Sponsor requests, PI must delete Sponsor confidential information before publication and/or delay publication for 60 days so Sponsor can file for patents or take other action to protect its patent rights.